CLINICAL TRIAL: NCT03237416
Title: A Phase I, Non-randomized, Open-label, Fixed-sequence Study to Investigate the Effect of Darolutamide (ODM-201) on the Pharmacokinetics of a Probe Substrate of CYP3A4 and P-gp in Healthy Male Volunteers
Brief Title: Drug-drug-interaction Study to Assess the Effect of Darolutamide on the Pharmacokinetics of Probe Substrates of CYP3A4 and P-gp in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Collaborators: Orion Corporation, Orion Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18860; 2017-001116-11 (EudraCT Number)
Record Dates: First submitted 2017-07-26; First posted 2017-08-02 (Actual); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Prostatic Neoplasms
Keywords: Drug-drug interaction
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Dabigatran; Midazolam; darolutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BAY1841788/Healthy subjects (Experimental): Period 1: intake of Midazolam and Dabigatran etexilate at day 1 followed by Period 2: intake of Darolutamide at days 1-11 (twice daily), intake of dabigatran etexilate at days 3 and 9, intake of Midazolam at day 9
  Interventions: Drug: Dabigatran etexilate; Drug: Midazolam; Drug: BAY1841788 (darolutamide)

INTERVENTIONS:
Drug: Dabigatran etexilate — In Period 1, Day 1 a single dose of 75 mg will be administered after breakfast In Period 2, Day 3 a single dose of 75 mg will be administered prior to breakfast In Period 2, Day 9 a single dose of 75 mg will be administered after breakfast
Drug: Midazolam — In Period 1, Day 1 a single dose of 1 mg will be administered after breakfast In Period 2, Day 9 a single dose of 1 mg will be administered after breakfast
Drug: BAY1841788 (darolutamide) — In Period 2, Days 1-11 600 mg twice a day (as 2 x 300 mg tablets) will be administered after breakfast

SUMMARY:
Evaluate the effect of darolutamide on the pharmacokinetics of a probe CYP3A4 substrate and Pgp substrate

ELIGIBILITY:
Inclusion Criteria:

* Healthy subject - as determined by the investigator or medically qualified designee based on medical evaluations including medical history, physical examination, laboratory tests and cardiac monitoring.
* Gender: Male.
* Age: 45 to 65 years (inclusive) at the screening visit.
* Race: White.
* Body mass index (BMI): ≥18.0 and ≤30.0 kg/m2.
* Agree to use condoms as an effective contraception barrier method and refrain from sperm donation during the whole study (starting after informed consent) and for 3 months after the end of treatment with darolutamide.

In addition, participants must agree to utilize a second reliable method of contraception simultaneously. The second method which has to be used by a female partner of childbearing potential can be one of the following methods: diaphragm or cervical cap with spermicide or intra-uterine device or hormone-based contraception. Therefore, contraception methods to be used by male subjects and female partners are in line with clinical trial facilitation group recommendations related to contraception in clinical trials.

* Ability to understand and follow study-related instructions.
* Results of alcohol tests are negative at screening and on Study Day -1.
* Confirmation of the subject's health insurance coverage prior to the first screening examination/visit.

Exclusion Criteria:

* Existing relevant diseases of vital organs (e.g. liver diseases, heart diseases), central nervous system (for example seizures) or other organs (e.g. diabetes mellitus).
* Incompletely cured pre-existing diseases for which it can be assumed that the absorption, distribution, metabolism, elimination and effects of the study drugs will not be normal.
* Known history of hypersensitivity (or known allergic reaction) to medications including any ingredient of midazolam, benzodiazepines, dabigatran etexilate, or darolutamide.
* Relevant hepatic disorders like cholestasis, disturbances of bilirubin metabolism, any progressive liver disease.
* Relevant renal disorders like recurrent glomerulonephritis, renal injury, and renal insufficiency. However, a history of a single episode of uncomplicated nephrolithiasis will not prevent participation.
* CYP3A4 inhibitors within 1 week or 5 drug half-lives, whichever is longer, before start of study treatment or during the study.
* CYP3A4 inducers as well as St John's Wort within 28 days or 5 drug half-lives, whichever is longer, before start of study treatment or during the study.
* Known BCRP and OATP substrates within 28 days or 5 drug half-lives, whichever is longer, before start of study treatment or during the study.
* P-gp inducers (e.g. rifampin) within 28 days or 5 drug half-lives, whichever is longer, before start of study treatment or during the study.
* P-gp inhibitors within 1 week or 5 drug half-lives, whichever is longer, before start of study treatment or during the study.

Ages: 45 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2017-10-05 (Actual); Study Completion 2017-12-18 (Actual)

PRIMARY OUTCOMES:
AUC in plasma of non-conjugated dabigatran (AUC(0-tlast), if AUC cannot be calculated) | Period 1, Day 1: Predose, and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 72 hours post dosing Period 2, Day 3 and 9: Predose, and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 72 hours post dosing
  Exposure of non-conjugated dabigatran in plasma following a single administration of dabigatran etexilate AUC: area under the concentration vs. time curve from zero to infinity after single (first) dose AUC(0-tlast): AUC from time 0 to the last data point > LLOQ
C(max) in plasma of non-conjugated dabigatran | Period 1, Day 1: Predose, and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 72 hours post dosing Period 2, Day 3 and 9: Predose, and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 72 hours post dosing
  Maximum plasma concentration of non-conjugated dabigatran in plasma following a single administration of dabigatran etexilate Cmax: maximum observed drug concentration in measured matrix after single dose administration
AUC in plasma of midazolam (AUC(0-tlast), if AUC cannot be calculated) | PPeriod 1, Day 1: Predose, and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 72 hours post dosing Period 2, Day 3 and 9: Predose, and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 72 hours post dosing
  Exposure of midazolam in plasma following a single administration of midazolam
C(max) in plasma of midazolam | Period 1, Day 1: Predose, and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 72 hours post dosing Period 2, Day 3 and 9: Predose, and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 72 hours post dosing
  Maximum plasma concentration of midazolam in plasma following a single administration of midazolam

SECONDARY OUTCOMES:
Number of subjects with study drug-related treatment-emergent Adverse Event (TEAE) | 30 days following last intake of Investigational Product
AUC in plasma of total dabigatran (AUC(0-tlast), if AUC cannot be calculated) | Period 1, Day 1: Predose, and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 72 hours post dosing Period 2, Day 3 and 9: Predose, and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 72 hours post dosing
  Exposure of total dabigatran in plasma following a single administration of dabigatran etexilate
C(max) in plasma of total dabigatran | Period 1, Day 1: Predose, and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 72 hours post dosing Period 2, Day 3 and 9: Predose, and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 72 hours post dosing
  Maximum plasma concentration of total dabigatran in plasma following a single administration of dabigatran etexilate
AUC in plasma of 1-OH midazolam (AUC(0-tlast), if AUC cannot be calculated) | Period 1, Day 1: Predose, and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 72 hours post dosing Period 2, Day 3 and 9: Predose, and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 72 hours post dosing
  Exposure of 1-OH midazolam in plasma following a single administration of midazolam
C(max) in plasma of 1-OH midazolam | PPeriod 1, Day 1: Predose, and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 72 hours post dosing Period 2, Day 3 and 9: Predose, and 0.25, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 10, 12, 15, 24, 36, 48, 72 hours post dosing
  Maximum plasma concentration of 1-OH midazolam in plasma following a single administration of midazolam

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- CRS Clinical-Research-Services Mannheim GmbH, Mannheim, Baden-Wurttemberg, Germany